CLINICAL TRIAL: NCT03012074
Title: From Episodic to Real-Time Care in Diabetes Self-Management
Brief Title: Episodic to Real-Time Care in Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00071569
Record Dates: First submitted 2016-12-21; First posted 2017-01-06 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type II
Keywords: diabetes, mHealth, mobile health technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Type II Diabetes (Experimental): Patients with Type II Diabetes
  Interventions: Behavioral: Type 2 Diabetes Self-Management

INTERVENTIONS:
Behavioral: Type 2 Diabetes Self-Management — Patients with Type 2 Diabetes

SUMMARY:
This study will use mobile health technologies to provide everyday data to help patients and their care providers better understand illness dynamics and develop adaptive approaches to improve health outcomes in diabetes. Specifically, the study will identify strategies to help patients adapt using multiple types of self-generated diabetes-related data and help providers guide patients to better self-manage in real-time, when guidance is needed most.

DETAILED DESCRIPTION:
The investigators will conduct a mixed-methods exploratory designed study and recruit 60 adult patients (age ≥ 18) with type 2 diabetes who will track relevant clinical data over 6 months. Participants will be asked to use a wireless glucose monitor, a cellular body scale, and a wrist-worn accelerometer, and respond to short bi-weekly text message-based surveys on medication adherence for 6 months. Data generated from the devices will be plotted as trajectories that will allow us to conduct trajectory analyses and identify missing data points and trends leading to attrition, in order to assess the feasibility of having patients engage in this type of self-monitoring for 6 months. A subset of 20 patients will be interviewed via telephone at the end of their 6 month self-monitoring period to discuss their adaptive challenges and successes over the study period. The investigators will present the trajectories of their data during patient interviews using a visual that we will e-mail or postal mail, depending on patient preference. This will facilitate discussion of the challenges participants face in self-management and adaptive practices participants use. Following the 6 months of self-monitoring, we will conduct interviews with health care providers in which the investigators will present the data trajectories and explore ways to achieve continual communication and address real-time challenges with diabetes self-management.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* able to speak and read English
* diagnosed with type 2 diabetes mellitus
* told by their primary care provider to monitor their blood sugar daily
* owning and using a smart phone
* capable of giving informed consent
* with no pre-existing severe medical condition(s) that would interfere with study participation (e.g., renal failure, severe orthopedic conditions or joint replacement scheduled within 6 months, paralysis, or cancer)

Exclusion Criteria:

* active dementia or psychiatric illness
* reside in a nursing home
* participating in another self-management study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with type II diabetes who adhere to using mobile technologies to self-monitor multiple types of diabetes-related data | 6 months

SECONDARY OUTCOMES:
Explore the adaptive challenges of patients self-managing diabetes, using monthly interviews over 6 months. | 6 months
Explore the successes of patients self-managing diabetes, using monthly interviews over 6 months. | 6 months
Change in daily blood glucose levels in patients with diabetes over a 6 month period | 6 months
  Data generated from the phone-tethered glucose monitor and plotted as a trajectory over a 6 month period
Change in daily weight in patients with diabetes over a 6 month period | 6 months
  Data generated from the cellular body scale and plotted as a trajectory over a 6 month period
Change in daily physical activity in patients with diabetes over a 6 month period | 6 months
  Data generated from the wrist-worn accelerometer and plotted as a trajectory over a 6 month period
Medication adherence Survey | 6 months
  bi-weekly text message-based surveys on medication adherence over a 6 month period.

OTHER OUTCOMES:
Explore health care providers' perspectives on using real-time data, by conducting one-time, individual interviews over a 2 month period. | 2 months
  Explore ways to achieve continual communication that addresses real-time challenges with diabetes self-management while presenting data trajectories during provider interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Shaw, PhD, RN, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No